CLINICAL TRIAL: NCT07265310
Title: Pre-therapeutic Value of Emergency Spine MRI in Patients With Thoraco-lumbar Spine Injuries - A Prospective Study.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Radio02
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Spinal Fracture; Spinal Injuries; Wounds and Injuries
MeSH Terms: conditions — Spinal Fractures; Spinal Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Clinical value of spine MRI in therapeutic management of patients admitted for thoraco-lumbar spine injuries, in addition to ct-scan. — Therapeutic possibilities include conservative, percutaneous and invasive (surgery) treatments. The aim of the study is to evaluate whether spine mri changes the therapeutic management.

SUMMARY:
The main objective is to determine whether the realisation of an emergency spine MRI in addition to CT-scan( Computed Tomography) in patients with thoraco-lumbar spine injuries changes the therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years old admitted in the emergency department for a thoracolumbar spine trauma, who have undergone a ct scan and a mri of the spine.

Exclusion Criteria:

* Underlying pathology of the spine, AO spine A0 and AO spine C traumas, neurological symptoms or clinical examination not done for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults admitted in the emergency departement of the university hospital of Nice, France.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in therapeutic management of thoraco-lumbar spine injuries | At the inclusion
  The Bowker test will be used to analyze paired categorical data and determine whether there is symmetry between the rows and columns of a square table (3x3; before/after MRI)

SECONDARY OUTCOMES:
Occult fractures | At the inclusion
  Account of fractures only viewed with MRI, defined as T1 hyposignal and T2 STIR (short TI inversion recovery .hypersignal of a vertebral endplate.
Change in AO spine classification | At the inclusion
  Comparison of CT scan and MRI AO spine classification of injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de France, Nice, Alpes Maritimes, France